CLINICAL TRIAL: NCT00790946
Title: Effects of Valsartan on Metabolic Syndrome in Patients With Hypertension
Brief Title: Kagoshima Collaborate Trial in Metabolic Syndrome (KACT Study)
Acronym: KACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kagoshima University (Other)
Responsible Party: Chuwa Tei / Professor, Kagoshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVM-RCT-2006-06
Record Dates: First submitted 2008-10-10; First posted 2008-11-14 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension; Obesity
Keywords: valsartan; Metabolic syndrome
MeSH Terms: conditions — Hypertension; Obesity; Metabolic Syndrome | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): Valsartan 80 to 160mg
  Interventions: Drug: Valsartan
- standard therapy (No Intervention)

INTERVENTIONS:
Drug: Valsartan — Valsartan 80 to 160 mg
  Arms: Valsartan

SUMMARY:
The purpose of this study is to consider the following points in patients with hypertension who complicated by metabolic syndrome for Valsartan basis treatment and an existing, standard treatment.

* Blood pressure control
* Changing of adiponectin and plasminogen activator inhibitor-1
* Influence metabolizing and cardiac function, etc.

DETAILED DESCRIPTION:
The primary endpoints are:

* blood pressure control
* Adiponectin and plasma type1 plasminogen active inhibitor

The secondary endpoints are

* HOMA-IR
* HbA1c
* TNF-α
* IL-6
* Plasma B-type natriuretic peptide
* LVMI
* E/A ratio
* Tei-index
* Apo-J

ELIGIBILITY:
Inclusion Criteria:

* Out patients with hypertension male and female
* Systolic blood pressure (SBP)≧140mmHg and/or diastolic blood pressure (DBP)≧90 mmHg
* Waist Surrounding diameter male≧85cm female≧90cm
* Patient who is treating either high triglyceride,low HDL,or diabetes mellitus
* Patient who is untreatment high triglyceride blood syndrome and low HDL blood syndrome,diabetes mellitus is triglceride≧150mg/dl and/or HDL cholesterol < 40 mg/dl or fasting blood glucose ≧110 mg/dl
* Untreated patients with hypertension,or patients is treated with antihypertensive agents except for ACE-I and ARB

Exclusion Criteria:

* Patient who is using ACE-I and ARB
* Serum creatinine ≧ 3 mg/dl
* Liver impairment
* History of allergy to valsartan
* Pregnant women
* Judgment by the physician that participation was unwise on the basis of patient characteristics and drug safety

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure, Adiponectin and PAI-1 concentration | 1 year

SECONDARY OUTCOMES:
HOMA-IR | 1 year
HbA1c | 1 year
TNF-α | １ year
IL-6 | 1 year
BNP | 1 year
LVMI | 1 year
E/A ratio | 1 year
Tei-index | 1 year
Apo-J | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chuwa Tei, MD, PhD, Study Chair — Department of Cardiovascular,Respiratory & Metabolic Medicine Granduate School of Medicine Kagoshima University
Locations (1):
- Chuwa Tei,MD,FACC,FAHA, Kagoshima, Kagoshima-ken, Japan

REFERENCES:
- [Derived] Miyata M, Ikeda Y, Nakamura S, Sasaki T, Abe S, Minagoe S, Torii H, Lee S, Tateishi S, Kihara K, Ohba I, Kajiya S, Furusho Y, Hamasaki S, Tei C; Kagoshima Collaborate Trial in Metabolic Syndrome (KACT-MetS) Investigators. Effects of valsartan on fibrinolysis in hypertensive patients with metabolic syndrome. Circ J. 2012;76(4):843-51. doi: 10.1253/circj.cj-12-0153. PMID 22451451